CLINICAL TRIAL: NCT03299010
Title: 10-year Risk Prediction Models of Complications and Mortality of Diabetes Mellitus in Chinese Patients in Primary Care in Hong Kong
Brief Title: 10-year Risk Prediction Models of Complications and Mortality of DM in Hong Kong
Status: Completed | Type: Observational
Sponsor: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Professor Cindy L.K. Lam, Head of Department, The University of Hong Kong
Other Study IDs: HKUCTR-2232
Record Dates: First submitted 2017-09-27; First posted 2017-10-02 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Diabetes Mellitus; Cardiovascular Diseases; Mortality; Primary Health Care
Keywords: Diabetes Mellitus; Risk; Complications; Mortality; Cardiovascular Diseases; Chinese; Prediction
MeSH Terms: conditions — Diabetes Mellitus; Cardiovascular Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- DM patient: Patients with a documented clinical diagnosis of DM and were receiving care in the Hospital Authority (HA) primary care General Out-Patient Clinics (GOPC) and Family Medicine Clinics (FMC) on or before 1 July 2006 identified from the HA clinical management system (CMS) database.

SUMMARY:
Diabetes Mellitus (DM) is a well-recognized public health issue worldwide. DM can lead to many complications resulting in morbidity and mortality, approximately 70% of DM related deaths were attributed to cardiovascular diseases (CVD).

Objectives:

To develop 10-year risk prediction models for CVD, end stage renal disease (ESRD) and all-cause mortality among Chinese patients with DM in primary care.

Hypotheses:

1. Patient socio-demographic, clinical parameters, disease characteristics and treatment modalities are predictive of 10-year risk of CVD, ESRD and all-cause mortality.
2. Risk prediction models developed from this study should have over 70% of discriminating power.

Design and Subjects:

10-year retrospective cohort study. All Chinese patients who were clinically diagnosed to have DM and were receiving care in the public (Hospital Authority) primary care clinics on or before 1 July 2006 will be followed up until 31 December 2016.

Main outcomes measures:

For total CVD, CHD, stroke, heart failure, ESRD, all-cause mortality

1. 10-year incidence;
2. Predictive factors

Data analysis:

Two thirds of subjects will be randomly selected as the training sample for model development. Cox regressions will be used to develop sex-specific 10-year risk prediction models for each outcome. The validity of models will be tested on the remaining one third of subjects by Harrell C statistics and ROC

Expected results:

Risk prediction models will enable accurate risk stratification and cost-effective interventions for Chinese DM patients in primary care.

DETAILED DESCRIPTION:
This study aims to develop 10-year risk prediction models for total CVD and all-cause mortality among Chinese diabetic patients in primary care. Risk prediction models for individual DM complications including CHD, heart failure, stroke and ESRD will also be developed.

The objectives are to:

1. Calculate the 10 years incidence of total CVD, all-cause mortality and each major DM complication in Chinese DM patients in primary care.
2. Determine the risk factors that significantly predict total CVD, all-cause mortality and each major DM complication for Chinese DM patients in primary care.
3. Develop and validate risk prediction models for total CVD, all-cause mortality and each major DM complication for Chinese DM patients in primary care.
4. Develop a risk prediction nomogram and chart for the risk of total CVD, all-cause mortality for Chinese DM patients in primary care

Hypotheses:

1. Patient socio-demographic, clinical parameters, disease characteristics, and treatment modalities are predictive of 10-year risk of total CVD, all-cause mortality and individual DM complication as a dependent variable.
2. The risk prediction models for total CVD, all-cause mortality and individual DM complication developed in this study can have over 70% of discriminating power.

ELIGIBILITY:
Inclusion Criteria:

1. At least 1 GOPC/FMC attendance on or within 1 year before 1 July 2006
2. Had a CMS (Clinical Management System) record in the Hospital Authority (HA) of the coding of ICPC-2 of T89 (Diabetes insulin dependent) or T90 (Diabetes non-insulin dependent) on or before 1 July 2006

Exclusion Criteria:

1. Patients who had a diagnosis of any DM complications defined by the relevant ICPC-2 or ICD-9-CM on or before 1 July 2006
2. Patients exclusively managed by Specialist Out-Patient Clinic (SOPC) on or before 1 July 2006.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The cohort will include all patients with a documented clinical diagnosis of DM and were receiving care in the Hospital Authority (HA) primary care General Out-Patient Clinics (GOPC) and Family Medicine Clinics (FMC) on or before 1 July 2006 identified from the HA clinical management system (CMS) database.
Sampling Method: Probability Sample
Enrollment: 141516 (Actual)
Dates: Start 2017-07-01 (Actual); Primary Completion 2018-12-31 (Actual); Study Completion 2019-12-31 (Actual)

PRIMARY OUTCOMES:
The incidence of total CVD, all-cause mortality and each of 4 major DM complications (CHD, stroke, heart failure and ESRD) over 10 years | 10 years
  Calculate the 10 years incidence of total CVD, all-cause mortality and each major DM complication in Chinese DM patients in primary care.
  CVD is defined as the presence of any of CHD, heart failure and stroke. CHD includes all ischaemic heart disease, myocardial infarction, coronary death or sudden death as indicated by the ICPC-2 K74 to K76 or ICD-9-CM 410.x, 411.x to 414.x, 798.x codes. Heart failure is defined by the ICPC-2 K77 or ICD-9-CM 428.x. Stoke (fatal and non-fatal stroke) is defined by the ICPC-2 K89 to K91 or ICD-9-CM 430.x to 438.x codes.
Factors predictive of total CVD, all-cause mortality and each of 4 major DM complications (CHD, stroke, heart failure and ESRD) over 10 years | 10 years
  Determine the risk factors that significantly predict total CVD, all-cause mortality and each major DM complication for Chinese DM patients in primary care.
10-year risk prediction models for total CVD, all-cause mortality and each of 4 major DM complications (CHD, stroke, heart failure and ESRD) | 10 years
  Develop and validate risk prediction models for total CVD, all-cause mortality and each major DM complication for Chinese DM patients in primary care.
Factors that have sufficient power to classify Chinese DM patients in primary care into risk group in terms of total CVD and all-cause mortality | 10 years
  Develop a risk prediction nomogram and chart for the risk of total CVD, all-cause mortality for Chinese DM patients in primary care

CONTACTS AND LOCATIONS:
Overall Officials: Cindy L.K. Lam, Principal Investigator — Department of Family Medicine and Primary Care, University of Hong Kong
Locations (2):
- Department of Family Medicine & Primary Care, University of Hong Kong, Hong Kong, Hong Kong, China
- The University of Hong Kong, Hong Kong, Hong Kong

REFERENCES:
- [Derived] Dong W, Fong DYT, Yoon JS, Wan EYF, Bedford LE, Tang EHM, Lam CLK. Generative adversarial networks for imputing missing data for big data clinical research. BMC Med Res Methodol. 2021 Apr 20;21(1):78. doi: 10.1186/s12874-021-01272-3. PMID 33879090
- [Derived] Wan EYF, Yu EYT, Chin WY, Fung CSC, Kwok RLP, Chao DVK, Chan KH, Hui EM, Tsui WWS, Tan KCB, Fong DYT, Lam CLK. Ten-year risk prediction models of complications and mortality of Chinese patients with diabetes mellitus in primary care in Hong Kong: a study protocol. BMJ Open. 2018 Oct 15;8(10):e023070. doi: 10.1136/bmjopen-2018-023070. PMID 30327405
- See also: Review on continuity of care on health outcomes in patients with DM/HT — https://doi.org/10.1186/s12875-021-01493-x
- See also: Continuity of care and complications in patients with HT — https://doi.org/10.3399/BJGP.2023.0150

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-03-04): https://cdn.clinicaltrials.gov/large-docs/10/NCT03299010/Prot_SAP_000.pdf